CLINICAL TRIAL: NCT04201925
Title: Objective and Subjective Functional Outcomes Following Upper Blepharoplasty
Brief Title: Functional Changes After Upper Blepharoplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, Lecturer of ophthalmology, Benha University
Other Study IDs: hamaky3
Record Dates: First submitted 2019-11-24; First posted 2019-12-17 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Eyelid Diseases
Keywords: blepharoplasty, visual field
MeSH Terms: conditions — Eyelid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- blepharoplasty: Patients will undergo blepharoplasty surgery
  Interventions: Procedure: upper blepharoplasty

INTERVENTIONS:
Procedure: upper blepharoplasty — excision of excess eyelid skin with or without strip of orbicularis muscle ; with or without upper orbital fat

SUMMARY:
Upper blepharoplasty is a common eyelid procedure. It associated with visual, cosmetic and functional changes .Investigator will evaluate outcome of this procedure.

DETAILED DESCRIPTION:
baseline and postoperative 1,3,6 and 12 months full ophthalmic examination was done.

Procedure is upper blepharoplasty.

ELIGIBILITY:
Inclusion Criteria:

• upper eyelid Dermatochalasis

Exclusion Criteria:

* Eyelid diseases
* previous eyelid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patient with upper eyelid Dermatochalasis and will undergo upper blepharoblasty procedure.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
visual field changes | 6 months
  Post operative visual field changes in form of change in visual field sensitivity decibel (dB)using Humphrey Field Analyzer( HFA) II-i (Carl Zeiss Meditec ,Jena, Germany)

SECONDARY OUTCOMES:
corneal topographic changes | 6 months
  Postoperative topographic changes of the cornea in form of central keratoconus index using Pentacam HR (Oculus GmbH, Wetzlar, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: TAREK R ELAHAMKY, MD, Principal Investigator — Benha university faculty of medicine
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates